CLINICAL TRIAL: NCT01314079
Title: Follow-up Study to Evaluate the Sustained Efficacy and Safety for the Patients With Adipoplus Injected in Phase II Clinical Trials(ANTG-ASC-202)
Brief Title: Follow-up Study of Autologous Cultured Adipose-derived Stem Cells for the Crohn's Fistula
Acronym: ANTG-ASC-203
Status: Completed | Type: Observational
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ANTG-ASC-203
Record Dates: First submitted 2011-03-08; First posted 2011-03-14 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2012-03

CONDITIONS: Crohn's Disease; Fistula
Keywords: Crohn's fistula; Autologous adipose derived stem cell
MeSH Terms: conditions — Crohn Disease; Fistula

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an open follow-up clinical trials to evaluate a sustained efficacy and safety of Adipoplus inj. for 10 months (12 months after final dose injection)after Phase II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* the patients who have participated in ANTG-ASC-202 clinical trial
* the patients who have experienced with Adipoplus in ANTG-ASC-202 trials
* the patients who submit written consents and is able to obey requirements of trials

Exclusion Criteria:

* pregnant or breast feeding
* autoimmune disease other than Crohn's disease
* infectious diseases including HBV, HCV or HIV
* who is not willing to use effective contraceptive methods during the study.
* active tuberculosis
* moderate to severe active or worsened Crohn's disease
* who have received Infliximab during or after ANTG-ASC-202 trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who have participated in phase II clinical trial (ANTG-ASC-202) and injected with Adipoplus at least once.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with Sustained efficacy of complete closure of fistula | Month 4, 10
  Proportion of patients whose fistula has been completely closed.

SECONDARY OUTCOMES:
Number of patients with sustained efficacy of closure of fistula | Month 2, 4, 10
  Proportion of patients with more than 50% closed of fistula (Month 2, 4, 10)
Number of patients with any adverse event | Month 2, 4, 10
  number of patients with any adverse event (Month 2, 4, 10)
Grade of Investigator's satisfaction | Month 2, 4, 10
  Grade of Investigator's satisfaction (Month 2, 4, 10)
  1. very satisfaction
  2. satisfacttion
  3. somewhat satisfaction
  4. unsatisfaction
  5. very unsatisfaction

CONTACTS AND LOCATIONS:
Overall Officials: CS You, MD, PhD, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - DaeHang Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul Asan Hospital, Seoul